CLINICAL TRIAL: NCT02142699
Title: Phase II Study of Heme Arginate in Patients Planned for Cardiac Surgery
Brief Title: Heme Arginate in Cardiac Surgery Patients
Acronym: HACS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Medical Research Council (Other Government); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SE01047; 2014-001021-32 (EudraCT Number)
Record Dates: First submitted 2014-05-09; First posted 2014-05-20 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Cardiac surgery; Ischaemia reperfusion injury; hemearginate
MeSH Terms: conditions — Acute Kidney Injury; Reperfusion Injury | interventions — heme arginate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heme arginate 1mg/kg (Active Comparator): This is the lower of the 2 doses of Heme arginate (HA). This will be given as a single dose of 1mg/kg on the first study visit.
  This is given over 1 hour intravenously.
  Interventions: Drug: Heme arginate
- Heme arginate 3mg/kg (Active Comparator): This is the larger dose, Heme arginate 3mg/kg (up to a maximum dose of 250mg)
  This will be given intravenously, as a single dose on the first study visit, over one hour.
  Interventions: Drug: Heme arginate

INTERVENTIONS:
Drug: Heme arginate
  Other Names: Normosang (Orphan Europe)

SUMMARY:
A recent analysis of over 4500 cardiac surgical patients at the Royal Infirmary of Edinburgh has confirmed that acute kidney injury (AKI) is not only a relatively common post-operative complication but is associated with prolonged hospital stay, and increased risk of death. There is currently no specific therapy available except supportive care.

In laboratory studies, heme arginate (HA), a drug licensed for human use, has been shown to upregulate the anti-inflammatory enzyme hemeoxygenase-1 (HO-1) and protect aged mice from acute kidney injury.

This study will bring this research into the human arena. It will aim to evaluate the minimum effective dose of HA and verify its safety in this specific group of patients. This will be the next step in investigating if HA could be a potential protective treatment for reducing AKI in patients about to have cardiac surgery.

Patients who are due to have cardiac surgery and are aged 60 or above will be approached for inclusion in the study. If agreeable, they will be randomly assigned to receive either HA at a dose of 1mg/kg or 3mg/kg. There will be 10 patients in each group.

Blood tests will be taken just before the study drug is given, at 6 hours, 24 hours and 7 days post dose. These samples will be used to examine the effect of HA on HO-1 at different doses, and will verify drug safety. Any adverse effects of the drug will be evaluated, although HA has an excellent safety profile when used as it is currently licensed for acute porphyria. Urine samples will also be collected to assess inflammation and quantify urinary biomarkers of AKI. This will set the scene for a randomised clinical trial of HA in cardiac surgical patients at high risk of AKI.

DETAILED DESCRIPTION:
AKI is a common condition which carries significant morbidity and mortality and has no current treatment except supportive care.

Cardiac surgery remains the standard of care for the revascularisation of the most severe coronary artery disease despite improvements in percutaneous coronary intervention. The nature of such surgery confers an ischaemic renal insult and it follows on that AKI is a relatively common complication. However, the reported incidence of AKI post cardiac surgery varies widely depending on the diagnostic criteria used. A recent retrospective analysis of 4572 cardiac surgical patients at the Royal Infirmary of Edinburgh over a 5 year period showed that 12.4% developed AKI by AKIN criteria post operatively. This was associated with an increased risk of death and prolonged inpatient stay.

Pre-clinical studies in murine models of ischaemia reperfusion injury (IRI) have demonstrated that the anti-inflammatory enzyme HO-1 is of interest as a potential target for therapeutic intervention. Heme arginate (HA) is a drug licensed for human use, as a treatment for acute porphyria. HA upregulates HO-1, and ameliorates IRI when given before injury in murine models of IRI. In Phase I clinical trials, HA has been shown to upregulate HO-1 and is well tolerated.

This is a single-blinded randomised trial of Heme arginate (HA) in patients who are due to have cardiac surgery. The aim of the study is to investigate the efficacy of HA in HO-1 upregulation and its safety in this patient cohort. This will inform a further clinical trial of HA as a preventative treatment for AKI in patients undergoing cardiac surgery.

Methods

Eligible patients will be those planned for elective cardiac surgery, identified at their Cardiothoracic outpatient clinic assessment, aged 60 or above.

HA (3mg/kg) upregulates HO-1 mRNA up to 2-fold at 24 hours post dose in healthy young volunteers. Power calculations based on an 80% power (at p<0.05) to detect at least 2 fold upregulation of HO-1 protein by western blot necessitate 2 groups of 10 (assuming standard deviation (SD) of ±1.5x). 20 patients will be recruited (10 per group).

Patients who agree to participate will be invited up for a study visit to the Clinical Research Facility at the Royal Infirmary of Edinburgh (RIE). If consent is given, participants will be randomised to receive HA at a dose of either 1 or 3mg/kg (maximum 250mg). Prior to the dose being given, routine observations (including blood pressure, pulse, respiratory rate, oxygen saturations and temperature) will be taken, and the trial team member will perform a routine examination of the cardiac and respiratory systems. An electrocardiogram (ecg) will be done for reference.

Blood samples to assess HO-1 expression in circulating monocytes will be taken prior to the administration of the study drug, and at 24 hours post dose. Samples for routine blood tests including full blood count (FBC), urea and electrolytes (U&E), C-reactive protein (CRP), liver function tests (LFT), and ferritin will be taken alongside those for monocyte isolation, with a further set on day 7. Serum (and urine) will be frozen for batch analysis and monocytes will be isolated by in-house protocols. Routine blood tests will be processed at the biochemistry and haematology laboratories at the RIE as per their usual methods.

Urine samples will be collected before the study drug is given, and at 24 hours and 7 days post dose. Urinalysis will be performed, and microalbuminuria and urinary biomarkers of tubular injury neutrophil gelatinase associated lipocalin(NGAL), interleukin 18(IL-18) & kidney injury molecule 1(KIM-1) will be quantified.

Routine clinical observations will be carried out for 6 hours post dose, at which time the patient will be allowed home in the absence of any adverse events. A second study visit at the Clinical Research Facility will be scheduled for 24 hours post dose (day 1), with a third study visit on day 7.

The second and third study visits will allow reporting of any adverse events, as well as an opportunity to perform routine observations and take further blood samples for HO-1 induction and in order to analyse safety.

All patients will be genotyped for the short or long repeat HO-1 promoter polymorphism (either homozygous or heterozygous) though this has not been shown to affect HO-1 induction by HA in previous studies.

The RIE cardiac surgery unit performs approximately 1000 cases per year, with just less than 80% aged 60 or over from our analysis of 4572 patients. A conservative estimate for time to meet recruitment to the study is 3 months.

ELIGIBILITY:
Inclusion Criteria:

Age ≥60

Planned for elective cardiac surgical procedure:

* Aortic valve replacement
* CABG

Exclusion Criteria:

Inability to give informed consent Hypersensitivity to HA Enrolment in other clinical trials Renal replacement therapy Planned for elective cardiac surgical procedure other than CABG or AVR (including combined CABG and AVR) Less than 2 weeks until planned cardiac surgery at time of study drug administration Active infection

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10-17 (Actual); Primary Completion 2015-10-16 (Actual); Study Completion 2015-11-16 (Actual)

PRIMARY OUTCOMES:
Upregulation of Heme oxygenase-1 protein expression in circulating monocytes | within 3 months of study completion

SECONDARY OUTCOMES:
Upregulation of heme oxygenase-1 messenger ribonucleic acid (mRNA) in circulating monocytes | within 3 months of completion
Urinary biomarkers of acute kidney injury | within 3 months of completion of study
  Samples will be collected pre dose and at 24 hrs and 7 days to determine the effect (if any) of Heme arginate on levels of urinary biomarkers of AKI in order to inform future interventional trials
Safety | at final study visit ie 7 days post dose (or at the resolution of any ongoing adverse event if this lasts longer than 7 days)
  This will be a composite outcome measure consisting of multiple routine measures of safety including adverse event reporting, and the biochemical and haematological data collected (eg renal function, liver function tests, full blood count)
Heme oxygenase-1 (HO-1) Genotype | within 3 months of study completion
  Patients will have their genotype for HO-1 gene recorded (for the long (L) or short (S) promoter region)- therefore they will be either LL, LS or SS. The study is not powered to detect any difference but will inform future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Hughes, MD, Principal Investigator — Professor of Experimental Nephrology, University of Edinburgh; David C Kluth, MD, Principal Investigator — Reader in Nephrology, University of Edinburgh; Vipin Zamvar, MD, Principal Investigator — Royal Infirmary of Edinburgh, NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom